CLINICAL TRIAL: NCT07385898
Title: Effect of Dexmedetomidine on Lung Protection in Elderly Patients Undergoing Laparoscopic Surgery for Colorectal Cancer
Acronym: Dex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: Research NO. 64 for 2023
Record Dates: First submitted 2023-12-13; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2023-04

CONDITIONS: Rectal Tumors; Tumor of Sigmoid Colon; Lung Injury; Surgery, Laparoscopic; Dexmedetomidine
MeSH Terms: conditions — Rectal Neoplasms; Sigmoid Neoplasms; Lung Injury | interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Experimental Group: Intravenous infusion of 1 μg/kg dexmedetomidine was initiated after induction of anesthesia and completed within 20 minutes, followed by a continuous infusion of 0.3 μg/kg/h until 30 minutes prior to the end of surgery. Control Group: An equivalent volume of normal saline was administered via the same method. Data was recorded at the corresponding time points.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): After anesthesia induction, intravenous infusion of dexmedetomidine at 1μg/kg was administered and completed within 20 minutes, followed by continuous infusion at 0.3μg/kg/h until 30 minutes prior to the end of surgery.
  Interventions: Drug: Dexmedetomidine
- Control (Placebo Comparator): After anesthesia induction, 0.25 ml/kg of normal saline was infused within 20 minutes, followed by a continuous infusion of 0.075 ml/kg/h until 30 minutes before the end of surgery.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — After anesthesia induction, intravenous infusion of dexmedetomidine at 1μg/kg was administered and completed within 20 minutes, followed by continuous infusion at 0.3μg/kg/h until 30 minutes prior to the end of surgery.
  Other Names: Dexmedetomidine Hydrochloride
  Arms: Dexmedetomidine
Other: Normal saline — After anesthesia induction, 0.25 ml/kg of normal saline was infused within 20 minutes, followed by a continuous infusion of 0.075 ml/kg/h until 30 minutes before the end of surgery.
  Other Names: Saline
  Arms: Control

SUMMARY:
The primary change in aging lung tissue among older people is atrophy, leading to a significant decline in ventilatory function. Intraoperative mechanical ventilation further decreases lung compliance and ventilatory function in elderly patients, making them more susceptible to respiratory dysfunction and postoperative pulmonary complications, which severely affects patient safety and postoperative recovery. Dexmedetomidine is a highly selective α2-adrenergic receptor agonist, and several studies have found that intravenous infusion of dexmedetomidine exerted lung protective effects during single-lung ventilation thoracic surgery. However, one study found that continuous intravenous dexmedetomidine infusion during low-temperature cardiac arrest aortic surgery did not improve perioperative respiratory mechanics and oxygenation. Therefore, this project aims to investigate the lung protective effects of continuous intravenous infusion of dexmedetomidine during laparoscopic surgery for elderly patients with rectal or sigmoid colon cancer.

DETAILED DESCRIPTION:
As the body ages, all organs and tissues gradually undergo aging. Research has found that aging becomes increasingly significant after age 60, with the main change in pulmonary tissue aging being atrophy and a substantial decrease in ventilatory function. In elderly patients undergoing surgery, mechanical ventilation during surgery further reduces lung compliance, leading to an increased risk of respiratory dysfunction and postoperative pulmonary complications, which severely affect patient safety and postoperative recovery. Furthermore, due to its advantages, such as minimal trauma, less postoperative pain, and faster wound recovery, laparoscopic surgery has gradually become an essential surgical approach. However, during surgery, pneumoperitoneum and head-down position can cause diaphragmatic elevation, increased thoracic pressure, increased airway pressure, decreased lung compliance, and further aggravation of respiratory dysfunction and postoperative pulmonary complications. Therefore, exploring effective measures to protect the lungs during the perioperative period has always been a critical research direction for anesthesiologists.

Dexmedetomidine is a highly selective α2-adrenergic receptor agonist that mainly functions as a sedative and hypnotic, often used as an adjuvant in anesthesia. In recent years, some studies have found that intravenous infusion of dexmedetomidine during single-lung ventilation in thoracic surgery can play a lung-protective role by reducing the inflammatory response, improving oxidative stress, improving respiratory mechanics, increasing oxygenation, and reducing postoperative pulmonary complications. In obese patients undergoing laparoscopic sleeve gastrectomy, continuous intravenous infusion of dexmedetomidine can improve respiratory mechanics and increase oxygenation. However, some studies have also found that constant intravenous infusion of dexmedetomidine during chest aortic surgery with low-temperature cardiac arrest does not improve perioperative respiratory mechanics and oxygenation. In addition, it is unclear whether dexmedetomidine also has a lung-protective effect in elderly patients undergoing laparoscopic surgery in the head-down position.

According to the latest data statistics, the incidence and mortality of colorectal cancer rank among the top five malignant tumors globally, making it one of the primary cancers that endanger life and health. Although colorectal cancer is showing a trend toward younger age, it is still predominantly seen in elderly patients. Laparoscopic surgery for tumor resection is the primary treatment method, and during the surgery, a head-down position is required to expose the surgical field fully. As the head-down angle is the same for rectal cancer and sigmoid colon cancer laparoscopic surgery, this project focuses on elderly patients undergoing laparoscopic rectal or sigmoid colon cancer surgery. It explores the lung-protective effect of continuous intravenous infusion of dexmedetomidine during surgery, providing guidance for anesthesia management in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective laparoscopic surgery for rectal or sigmoid colon cancer.
2. American Society of Anesthesiologists (ASA) physical status classification I-III.
3. Age ≥60 years and <85 years.
4. Voluntary participation and ability to understand and sign the informed consent form.

Exclusion Criteria:

1. Patients with obesity (BMI>28 kg/m2)
2. Grade 3 hypertensive patients (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg)
3. Patients with acute coronary syndrome, sinus bradycardia (heart rate <45 beats/minute), II or III degree atrioventricular block, or NYHA heart failure class III or IV
4. Patients with a history of severe chronic obstructive pulmonary disease (COPD) (GOLD stage III or IV), severe or uncontrolled bronchial asthma, lung infections, bronchiectasis, thoracic deformities, and chest diseases (such as mediastinal tumors and thoracic tumors)
5. Pulmonary artery pressure ≥ 60 mmHg
6. Patients with Child-Pugh Class B or C liver function
7. Patients with stage 4 or 5 chronic kidney disease
8. Patients with hyperthyroidism, pheochromocytoma
9. Patients with hearing, intellectual, communication, or cognitive impairments
10. Patients who cannot cooperate with the study for any reason, or whom the investigator deems unsuitable for inclusion in this trial.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-02-03 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
oxygenation index | When patients enter the operation room (T0), 5 minutes after completion of pneumoperitoneum and trendelenburg position (T1), 30 (T2) and 60 (T3) minutes after trendelenburg position, when extubate the endotracheal tube (about 30 min postoperatively, T4)
  oxygenation index is the ratio of partial pressure of O2 in arterial blood to fraction of inspired oxygen, namely PaO2/FiO2 ratio.

SECONDARY OUTCOMES:
PaCO2 | When patients enter the operation room (T0), 5 minutes after completion of pneumoperitoneum and trendelenburg position (T1), 30 (T2) and 60 (T3) minutes after trendelenburg position, when extubate the endotracheal tube (about 30 min postoperatively, T4)
  arterial carbon dioxide pressure assessed by arterial blood gas measurement.
EtCO2 | 5 minutes after establishment of pneumoperitoneum and trendelenburg position (T1), 30 minutes after trendelenburg position (T2), 60 minutes after trendelenburg position (T3)
  end-tidal carbon dioxide pressure assessed by arterial blood gas measurement.
Pplat | 5 minutes after establishment of pneumoperitoneum and trendelenburg position (T1), 30 minutes after trendelenburg position (T2), 60 minutes after trendelenburg position (T3)
  plateau pressure (Pplat) is the end-inspiratory airway pressure and is measured just after airflow has ceased, which is displayed automatically on the anesthesia machine.
Ppeak | 5 minutes after establishment of pneumoperitoneum and trendelenburg position (T1), 30 minutes after trendelenburg position (T2), 60 minutes after trendelenburg position (T3)
  peak airway pressure is the highest pressure measured during the respiratory cycle and is a function of both the resistance of the airways and the compliance of the respiratory system, which is displayed automatically on the anesthesia machine.
lung compliance | 5 minutes after establishment of pneumoperitoneum and trendelenburg position (T1), 30 minutes after trendelenburg position (T2), 60 minutes after trendelenburg position (T3)
  lung compliance is defined as the change in lung volume for a unit change in transalveolar pressure, which is displayed automatically on the anesthesia machine.
Vd/Vt | 5 minutes after establishment of pneumoperitoneum and trendelenburg position (T1), 30 minutes after trendelenburg position (T2), 60 minutes after trendelenburg position (T3)
  Vd/Vt represents dead space ventilation, which is the volume of ventilated air that does not participate in gas exchange. Vd/Vt = 1.14 × (PaCO2-EtCO2) / PaCO2-0.005.
Qs/Qt | When patients enter the operation room (T0), 5 minutes after completion of pneumoperitoneum and trendelenburg position (T1), 30 (T2) and 60 (T3) minutes after trendelenburg position, when extubate the endotracheal tube (about 30 min postoperatively, T4)
  Qs/Qt is a measurement of pulmonary shunt. It describes the percentage of blood that reaches the left side of the heart without picking up oxygen. Qs/Qt = (CcO2 - CaO2) / (CcO2 - CvO2), where CcO2 = pulmonary end-capillary O2 content, same as alveolar O2 content, CaO2 = arterial O2 content, CvO2 = mixed venous O2 content.
PA-aO2 | When patients enter the operation room (T0), 5 minutes after completion of pneumoperitoneum and trendelenburg position (T1), 30 (T2) and 60 (T3) minutes after trendelenburg position, when extubate the endotracheal tube (about 30 min postoperatively, T4)
  alveolar-arterial oxygen gradient measures the difference between the oxygen concentration in the alveoli and arterial system, which can be obtained from the arterial blood gas measurement.
SPO2 | When patients enter the operation room (T0), 5 minutes after trendelenburg position (T1), 30 (T2) and 60 (T3) minutes after trendelenburg position, when extubate the endotracheal tube (about 30 min postoperatively, T4), postoperative day 1-3
  oxygen saturation refers to the amount of oxygen bound to hemoglobin in arterial blood.
Blood pressure | When patients enter the operation room (T0), 5 minutes after trendelenburg position (T1), 30 (T2) and 60 (T3) minutes after trendelenburg position, when extubate the endotracheal tube (about 30 min postoperatively, T4), postoperative day 1-3
  Systolic blood pressure, diastolic blood pressure, mean arterial pressure
HR | When patients enter the operation room (T0), 5 minutes after trendelenburg position (T1), 30 (T2) and 60 (T3) minutes after trendelenburg position, when extubate the endotracheal tube (about 30 min postoperatively, T4), postoperative day 1-3
  hear rate
Lac | When patients enter the operation room (T0), 5 (T1), 30 (T2) and 60 (T3) min after trendelenburg position, and when the tracheal tube was extubated (T4)
  lactic acid in blood
WBC | before surgery, postoperative day 1
  White blood cell counting in blood
NEU | before surgery, postoperative day 1
  neutrophil counting in blood
NEU(%) | before surgery, postoperative day 1
  percentage of neutrophil in blood
TV | before surgery, postoperative day 1
  Tidal Volume
MVV | before surgery, postoperative day 1
  minute ventilation volume
RR | before surgery, postoperative day 1
  respiration rate
Postoperative pulmonary complications | postoperative day 1, 2, and 3
  The incidence of postoperative pulmonary complications was assessed according to the Assess Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) definition.
The length of postoperative hospital stay | From the first day after surgery until the date of discharged from the hospital, assessed up to 1 months.
  The days stayed in hosptial after surgery
Postoperative hospitalization costs | From the first day after surgery until the date of discharged from the hospital, assessed up to 1 months.
  All fees cost postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: ling Dan, BD, Principal Investigator — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available with the corresponding author when required.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available when published and kept for 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Jiang H, Kang Y, Ge C, Zhang Z, Xie Y. One-lung ventilation patients: Clinical context of administration of different doses of dexmedetomidine. J Med Biochem. 2022 Apr 8;41(2):230-237. doi: 10.5937/jomb0-33870. PMID 35510198
- [Background] Jannu V, Dhorigol MG. Effect of Intraoperative Dexmedetomidine on Postoperative Pain and Pulmonary Function Following Video-assisted Thoracoscopic Surgery. Anesth Essays Res. 2020 Jan-Mar;14(1):68-71. doi: 10.4103/aer.AER_9_20. Epub 2020 Mar 16. PMID 32843795
- [Background] Kostroglou A, Kapetanakis EI, Matsota P, Tomos P, Kostopanagiotou K, Tomos I, Siristatidis C, Papapanou M, Sidiropoulou T. Monitored Anesthesia Care with Dexmedetomidine Supplemented by Midazolam/Fentanyl versus Midazolam/Fentanyl Alone in Patients Undergoing Pleuroscopy: Effect on Oxygenation and Respiratory Function. J Clin Med. 2021 Aug 9;10(16):3510. doi: 10.3390/jcm10163510. PMID 34441805
- [Background] Lee SH, Kim N, Lee CY, Ban MG, Oh YJ. Effects of dexmedetomidine on oxygenation and lung mechanics in patients with moderate chronic obstructive pulmonary disease undergoing lung cancer surgery: A randomised double-blinded trial. Eur J Anaesthesiol. 2016 Apr;33(4):275-82. doi: 10.1097/EJA.0000000000000405. PMID 26716866
- [Background] Xia R, Xu J, Yin H, Wu H, Xia Z, Zhou D, Xia ZY, Zhang L, Li H, Xiao X. Intravenous Infusion of Dexmedetomidine Combined Isoflurane Inhalation Reduces Oxidative Stress and Potentiates Hypoxia Pulmonary Vasoconstriction during One-Lung Ventilation in Patients. Mediators Inflamm. 2015;2015:238041. doi: 10.1155/2015/238041. Epub 2015 Jul 26. PMID 26273134
- [Background] Hasanin A, Taha K, Abdelhamid B, Abougabal A, Elsayad M, Refaie A, Amin S, Wahba S, Omar H, Kamel MM, Abdelwahab Y, Amin SM. Evaluation of the effects of dexmedetomidine infusion on oxygenation and lung mechanics in morbidly obese patients with restrictive lung disease. BMC Anesthesiol. 2018 Aug 14;18(1):104. doi: 10.1186/s12871-018-0572-y. PMID 30103679
- [Background] Kim S, Park SJ, Nam SB, Song SW, Han Y, Ko S, Song Y. Pulmonary effects of dexmedetomidine infusion in thoracic aortic surgery under hypothermic circulatory arrest: a randomized placebo-controlled trial. Sci Rep. 2021 May 26;11(1):10975. doi: 10.1038/s41598-021-90210-w. PMID 34040043